CLINICAL TRIAL: NCT01957943
Title: Impact of Pre-treatment of Living-donor Liver Transplant Recipients With Omega 3 Enriched Lipid Emulsions on Graft and Patient Outcome. A Prospective, Randomized, Multi-central Trial.
Brief Title: Omega 3 Lipid Emulsions and Liver Transplantation
Acronym: OTLT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Yassen, Professor Doctor Amr M. Yassen, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LTX_SMOF_PRE_Eg
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2016-07

CONDITIONS: Ischemia Re-perfusion Injury
Keywords: Omega 3 lipid emulsions; Liver transplantation; Ischemia reperfusion injury; graft function
MeSH Terms: conditions — Reperfusion Injury | interventions — SMOFlipid; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): 38 patients Will receive standard oral diet 3 days before the operation will receive similar volume of 10% glucose solution Will receive same solution for 5 days postoperatively
  Interventions: Dietary Supplement: equivalent volume of 10% glucose solution
- OMEGA_PRE (Active Comparator): 38 patients Will receive standard oral diet 3 days before the operation will receive lipid supplementation 2 days before the operation with omega 3 enriched lipid emulsion (SMOFlipid) Will receive omega 3 enriched lipid emulsion (SMOFlipid) supplementation for 5 days postoperatively
  Interventions: Dietary Supplement: SMOFLipid
- OMEGA_POST (Active Comparator): 38 patients Will receive standard oral diet 3 days before the operation will receive glucose 10% solution 2 days before the operation Will receive omega 3 enriched lipid emulsion (SMOFlipid 20%) supplementation for 5 days postoperatively
  Interventions: Dietary Supplement: SMOFLipid

INTERVENTIONS:
Dietary Supplement: SMOFLipid
  Other Names: Omega 3 lipid emulsions
  Arms: OMEGA_POST; OMEGA_PRE
Dietary Supplement: equivalent volume of 10% glucose solution — Patients will receive same dose of 10% glucose solution for 2 days pre operatives and 5 days post-operative
  Other Names: control group
  Arms: Control

SUMMARY:
The study Aims to investigate the possible beneficial impact of peri-operative or post-operative administration of Omega 3 enriched lipid emulsions on recipients for living donor liver transplantation.

DETAILED DESCRIPTION:
Patients will be divided intro three groups, A control group will receive equivalent volume of glucose 10% solution both 3 days before and 5 days after the operation .

A peri-operative groups, in which patients will receive omega 3 enriched lipid emulsion (SMOFLipid) for 2 days pre-transplantation and 5 days post-transplantation A Post-operative group, in which patients will receive glucose 10% 3 days before the operation and omega 3 enriched lipid emulsion (SMOFLipid) for 5 days post-transplantation The primary outcome objective will be the incidence of Ischemia re-perfusion injury, secondary outcomes includes post-operative complications, graft and patient's outcomes and graft regeneration

ELIGIBILITY:
Inclusion Criteria:

* All liver transplant recipients

Exclusion Criteria:

* Budd chiari
* Previous upper abdominal surgery
* Re-transplantation
* Known allergy to the study emulsion

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Ischemia reperfusion injury | 5 days

SECONDARY OUTCOMES:
Liver functions | 5 days
Early graft regeneration | one month
  assessment of percent of liver regeneration 1 month PO
Late graft regeneration | 3 month
  assessment of percent of liver regeneration 13 months PO

OTHER OUTCOMES:
mortality | 28 days
Renal functions | 28 days
Infection | 28 days
length of hospital stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Yassen, MD, Study Chair — Mansoura University
Locations (1):
- Liver transplantation program - Gastroenterology surgical center - Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt